CLINICAL TRIAL: NCT04707794
Title: The Incidence, Risk Factors and Outcome of Postoperative Delirium in Elderly Patients Undergoing Non-cardiac Surgery: a Prospective Observational Study
Brief Title: Incidence of Postoperative Delirium in Elderly Patients Undergoing Non-cardiac Surgery
Status: Recruiting | Type: Observational
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Nitin Sethi, DNB, Senior Consultant & Associate Professor, Sir Ganga Ram Hospital
Other Study IDs: EC/12/20/1763
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly: Patients > 65 years age undergoing non-cardiac surgery will be administered general anesthesia maintained with sevoflurane or desflurane titrated to maintain anaesthesia depth of 50 (BIS score) using bispectral (BIS) index monitioring
  Interventions: Drug: Sevoflurane; Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane delivery will will be titrated to maintain anaesthesia depth of 50 (BIS score) using bispectral (BIS) index monitioring
Drug: Desflurane — Desflurane delivery will be titrated to maintain anaesthesia depth of 50 (BIS score) using bispectral (BIS) index monitioring

SUMMARY:
Postoperative delirium (POD) is the most common adverse neurologic complication that can occur in patients of any age. Its incidence varies across age groups and is substantially influenced by patient-related risk factors. POD occurs in 17%-61% of major surgical procedures. Several risk factors which contribute to the development of POD include age more than 60 years, pre-existing cognitive dysfunction, presence of comorbidities, sensorial deficits, malnutrition, polypharmacy, impaired physical mobility and frailty. Postoperative delirium has several wide ranging and adverse outcomes that are consistently associated with delirium such as mortality, increased length of hospital stay, and increased hospital costs. A recently devised tool for rapid assessment of delirium is the 4 A's test. It has now been validated for identifying delirium in the surgical population. The proposed prospective observational study will be conducted on 150 patients belonging to ASA Physical Status I-III of either sex, scheduled to undergo non-cardiac surgery under general anaesthesia (GA), requiring at least 24 hours of postoperative inpatient care. This prospective, observational study aims to evaluate the incidence, risk factors and outcomes of postoperative delirium in elderly patients more than 65 years of age undergoing non-cardiac surgery.

DETAILED DESCRIPTION:
The incidence of postoperative delirium (POD) following major surgery ranges from 17% to 61%.POD is the most frequent neurological complication that can occur in both the young and old, and its rate is considerably impacted by patient-related risk issues. The elderly population is believed to be more susceptible to POD, by virtue of being host to conditions such as a variety of comorbidities, malnutrition, concurrent cognitive dysfunction, frailty, sensorial and functional deficits, and polypharmacy.

Risk factors for delirium may be further identified as predisposing factors and precipitating factors. Predisposing factors are those that are present on admission and are not changeable, e.g. age, number and severity of co-morbid medical conditions, sensory impairment, history of cognitive impairment, sleep deprivation, immobility, and dehydration.Precipitating factors are those that trigger delirium while the patient is hospitalized. These may be infections, constipation, bladder catheterisation, procedures involving instrumentation, immobility, and sensory impairment

Postoperative delirium, especially in the elderly, significantly compromises patient recovery and imposes a heavy toll on patient well-being and the healthcare system. Postoperative delirium has several wide-ranging and adverse outcomes associated with it, such as mortality, increased length of hospital stay and increased hospital costs.

Several tools have been developed to track changes in mental status that could point to the onset of delirium. Among the tools employed for this purpose are the Sedation Scale, the Nursing-Delirium Screening Scale (Nu-DESC), and the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU).

However, there is a lack of consensus on the use of an appropriate tool to evaluate delirium in the postoperative period. The 4A's test is a screening instrument that has been designed for rapid and initial assessment of delirium. It has the added advantage of evaluating not only delirium but also postoperative cognitive dysfunction (POCD) which is the second most common complication in elderly surgical patients.

Delirium is a condition that is presumed to be avoidable in 30%-40% of cases which emphasizes the importance of attention to primary prevention.5 After the onset of delirium, little can be done to influence its duration, severity, or the possibility of recurrence. Thus, the necessity for identifying those at risk of developing postoperative delirium. It is imperative that hospitals should implement multimodal non-pharmacologic delirium prevention methods to identify and monitor patients at risk of developing this morbid condition.

There has been scant research in the developing world, including India in the sphere of postoperative delirium, a condition germane to practically all medical specialities and especially in the elderly population. Our study will research POD we expect to obtain evidence that will find the clinical application.

Our study will be focused on evaluating the incidence of POD in the elderly who will be posted for non-cardiac surgical procedures. We will also assess the association of postoperative delirium with risk factors such as frailty, cognitive dysfunction, impaired functional status, presence of comorbidities and polypharmacy. Other postoperative adverse events such as sedation, pain, postoperative nausea and vomiting will be recorded. Patient's length of stay in the hospital (LOS), any unanticipated ICU admission and mortality within 30 days will also be noted.

The following parameters will be recorded in all the patients,

1. Postoperative delirium: It will be evaluated using 4 A's test, three times in the first 24 hours postoperatively. A score of 0 suggests absence of delirium or severe cognitive impairment, score 1-3 suggests presence of possible cognitive impairment, and a score > 4 suggests the presence of delirium/ cognitive impairment.
2. Frailty: All eligible patients will be assessed preoperatively using the 9-point CFS. Score varies from 1-9 with fitness level very fit to terminally ill as depicted in the table
3. Cognitive dysfunction: Preoperative cognition will be assessed using the 5-point Mini-cog test. A score < 4 will be taken as cut-off for impaired cognitive function
4. Impaired physical mobility: All preoperative mobile patients will be subjected to Timed Up and Go (TUG) test. A score of <10 s is normal and score of <20 s need assistance.
5. Intraoperative hemodynamics (pulse, systolic blood pressure, diastolic blood pressure, and mean arterial blood pressure) will be recorded every 5-minutes intraoperatively and every 15-minutes postoperatively in the postoperative care unit (PACU) till discharge. A mean arterial blood pressure <65 mmHg persisting for greater than 5-minutes despite treatment will be defined as an episode of intraoperative hypotension.
6. Postoperative sedation:Sedation will be assessed postoperatively using the Richmond Agitation and Sedation Scale. Score varies from +4 to -5 and patient will be categorised from combative to unarousable as depicted in table.
7. Postoperative pain will be assessed using the 10-point Numeric Rating Scale (NRS)
8. Postoperative nausea and vomiting (PONV) It will be assessed using 3-point Likert scale (0- no nausea and vomiting, 1- nausea only, 2- vomiting)
9. Length of stay in the hospital and any unanticipated ICU admission will be noted.
10. All patients will be followed up postoperatively for 30-days and any occurrence of mortality will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age >65yrs
* Either sex
* ASA physical status I - III
* Elective non-cardiac surgical procedures under general anesthesia
* Clinical Frailty Score (CFS): 1-8
* Patients requiring at least 24 hours of postoperative inpatient care.

Exclusion Criteria:

* Clinical Frailty Score (CFS) of 9
* Patients diagnosed with dementia, severe psychiatric or neurological diseases
* Recent surgery within past 3-months
* History of recent head injury in the preceding 3 months
* Patients with uncompensated cardiovascular disease, hepato-renal insufficiency and uncontrolled endocrine disease
* Patients on anti-depressant, anti-anxiety, anti-convulsant and anti-parkinsonism medications
* Preoperative haemoglobin < 8 gm % and serum albumin < 3.5mg/dl
* Patient inability to give informed consent
* Presence of preoperative delirium as assessed by 4A'S Test (score ≥ 4)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients greater then 65 years age undergoing elective non-cardiac surgical procedures under general anesthesia
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | From end of surgery till 24 hours postoperatively
  Postoperative delirium will be assessed using 4 A's test.A score of 0 suggests absence of delirium or severe cognitive impairment, score 1-3 suggests presence of possible cognitive impairment, and a score > 4 suggests the presence of delirium/ cognitive impairment

SECONDARY OUTCOMES:
Postoperative Sedation | From end of surgery till 24 hours postoperatively
  Postoperative sedation will be assessed using the 10 point Richmond Agitation and Sedation Scale. +4 suggests overtly combative & violent, 0 suggests awake & quiet, and -5 suggets no response to voice or physical stimulation
Postoperative Pain | From end of surgery till 24 hours postoperatively
  It will be assessed using the 10-point Numeric Rating Scale (NRS). A score of 0 suggests 'no pain'and score of 10 suggests 'maximum pain'experienced
Postoperative nausea and vomiting | From end of surgery till 24 hours postoperatively
  It will be assessed using 3-point likert scale. A score of 0 suggests 'no nausea & vomiting'and a scoe of 2 suggests 'nausea & vomiting present'
Length of hospital stay | From end of surgery till discharge from the hospital
  The number of days the patient stays in the hospital post surgery till discharge will be recorded.
Unanticipated intensive care unit (ICU) admission | From end of surgery till 30 days postoperatively
  Any postoperative event necessitating ICU admission will be recorded
Mortality | From end of surgery till 30 days postoperatively
  Any mortality occurring within 30 days of surgery will be recorded

OTHER OUTCOMES:
Correlation of risk factors with postoperative delirium | From end of surgery till 24 hours postoperatively
  Correlation between age more than 75 years, frailty, cognitive dysfunction, impaired physical mobility, comorbidity and polypharmacy with postoperative delirium will be assessed using multivariate or univariate analysis as applicable

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Sethi, MBBS, DNB, Principal Investigator — Sir Ganga Ram Hospital; Bimla Sharma, MBBS, DGO, MD, FICA, MHA, Study Chair — Sir Ganga Ram Hospital; Chand Sahai, MBBS, DA, MD, Principal Investigator — Sir Ganga Ram Hospital; Jayashree Sood, MBBS, MD, FFRCA, PGDHHM, FICA, Study Director — Sir Ganga Ram Hospital
Locations (2):
- India (2):
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Sir Ganga Ram Hospital, New Delhi

IPD SHARING:
Plan to Share IPD: No